CLINICAL TRIAL: NCT00331019
Title: Rapid Detection of Group B Streptococcus Using a Bedside Microfluidics Device: 35-37 Week Study
Brief Title: Rapid Detection of Group B Strep- 35-37 Week Study
Status: Withdrawn | Type: Observational
Why Stopped: HandyLab device determined to not work for the science
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Mark Pearlman, S Jan Behrman Collegiate Professor of Reproductive Medicine, Professor of Obstetrics and Gynecology and Professor of Surgery, Medical School, University of Michigan
Other Study IDs: HandyLab #VVP00056
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Group B Streptococcus Neonatal Sepsis
Keywords: Streptococcus Group B; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether a rapid bedside diagnosis of Group B Strep growing in the vagina and rectum can be performed with similar success to the routine culture.

DETAILED DESCRIPTION:
Early Onset Group B Strep (GBS) neonatal infections is one of the leading infections in newborns, nearly all of which are acquired by vertical transmission at the time of childbirth. Most cases can be prevented by identifying women who are colonized with GBS in the vaginal-rectal area and giving these colonized women prophylactic antibiotics in labor. About 15 -20% of women are colonized and nearly all of these women are asymptomatic. Because it takes up to 48 hours to obtain culture results, it is currently recommended to perform cultures in the clinic about 3 - 5 weeks prior to their due date and then prophylaxing those women colonized with GBS with antibiotics when they come in to labor. There are several downsides to this strategy. All women who present with preterm labor are treated until culture results become available (overtreatment), women who go into labor while waiting for culture results are all treated (overtreatment), prior studies have shown 33% of women are positive at 35 weeks, but negative at birth (overtreatment) and 10% are negative at 35 weeks and positive at birth (undertreatment), lost or missing culture results (over- or undertreatment). Using microfluidics and fluorescent PCR, a new test can identify GBS reliably in 30 to 45 minutes in vitro. This study proposes to evaluate the clinical performance (sensitivity, specificity, positive and negative predictive value) of the microfluidic rapid GBS technique in selected women presenting at 35 - 37 weeks to antenatal clinics at the University of Michigan compared to standard culture.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older
* Mentally capable of giving informed consent
* Presentation for regularly scheduled 35-37 week cultures

Exclusion Criteria:

* Inability to give informed consent
* Evidence of ruptured membranes by clinical or laboratory criteria
* Use of any antibiotic within the previous 7 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older who present for prenatal cultures in clinic at 35-37 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Pearlman, MD, Principal Investigator — University of Michigan, Obstetrics & Gynecology
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Boyer KM, Gotoff SP. Prevention of early-onset neonatal group B streptococcal disease with selective intrapartum chemoprophylaxis. N Engl J Med. 1986 Jun 26;314(26):1665-9. doi: 10.1056/NEJM198606263142603. PMID 3520319
- [Background] Yancey MK, Schuchat A, Brown LK, Ventura VL, Markenson GR. The accuracy of late antenatal screening cultures in predicting genital group B streptococcal colonization at delivery. Obstet Gynecol. 1996 Nov;88(5):811-5. doi: 10.1016/0029-7844(96)00320-1. PMID 8885919
- [Background] Schrag S, Gorwitz R, Fultz-Butts K, Schuchat A. Prevention of perinatal group B streptococcal disease. Revised guidelines from CDC. MMWR Recomm Rep. 2002 Aug 16;51(RR-11):1-22. PMID 12211284
- [Background] Edwards RK, Clark P, Duff P. Intrapartum antibiotic prophylaxis 2: positive predictive value of antenatal group B streptococci cultures and antibiotic susceptibility of clinical isolates. Obstet Gynecol. 2002 Sep;100(3):540-4. doi: 10.1016/s0029-7844(02)02097-5. PMID 12220775
- [Background] ACOG committee opinion. Prevention of early-onset group B streptococcal disease in newborns. Number 173--June 1996. Committee on Obstetric Practice. American College of Obstetrics and Gynecologists. Int J Gynaecol Obstet. 1996 Aug;54(2):197-205. No abstract available. PMID 9236325
- [Background] Centers for Disease Control and Prevention (CDC). Laboratory practices for prenatal Group B streptococcal screening and reporting--Connecticut, Georgia, and Minnesota, 1997-1998. MMWR Morb Mortal Wkly Rep. 1999 May 28;48(20):426-8. PMID 10365633
- [Background] Centers for Disease Control and Prevention (CDC). Adoption of hospital policies for prevention of perinatal group B streptococcal disease--United States, 1997. MMWR Morb Mortal Wkly Rep. 1998 Aug 21;47(32):665-70. PMID 9729032
- [Background] Yancey MK, Armer T, Clark P, Duff P. Assessment of rapid identification tests for genital carriage of group B streptococci. Obstet Gynecol. 1992 Dec;80(6):1038-47. PMID 1448249
- [Background] Walker CK, Crombleholme WR, Ohm-Smith MJ, Sweet RL. Comparison of rapid tests for detection of group B streptococcal colonization. Am J Perinatol. 1992 Jul;9(4):304-8. doi: 10.1055/s-2007-999247. PMID 1627226
- [Background] Bergeron MG, Ke D, Menard C, Picard FJ, Gagnon M, Bernier M, Ouellette M, Roy PH, Marcoux S, Fraser WD. Rapid detection of group B streptococci in pregnant women at delivery. N Engl J Med. 2000 Jul 20;343(3):175-9. doi: 10.1056/NEJM200007203430303. PMID 10900276